CLINICAL TRIAL: NCT01000324
Title: An Open Single Centre Study to Evaluate the Long-term Antibody Persistence and Immune Memory Between 16 and 20 Years After the Primary Study HAB-028 (208127/021) in Which Healthy Adults Were Vaccinated With Twinrix Adult Following a Three-dose Schedule.
Brief Title: Antibody Persistence & Immune Memory in Healthy Adults Previously Vaccinated With Twinrix Adult
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112267
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis A; Hepatitis B
Keywords: Hepatitis A; Hepatitis B
MeSH Terms: conditions — Hepatitis A; Hepatitis B | interventions — Blood Specimen Collection; Engerix-B; Hepatitis A Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Twinrix Group (Experimental): Pooled group of subjects from groups who were vaccinated with either Lot 1, Lot 2 or Lot 3 of Twinrix in the primary study according to a 0, 1, 6-Month schedule
  Interventions: Procedure: Blood sampling; Biological: Engerix-B; Biological: Havrix

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling at Year 16, 17, 18, 19 and 20 and at the time of challenge dose administration and 14 days and one month after challenge dose administration (if challenge dose needed).
Biological: Engerix-B — Engerix-B will be administered to subjects who are not seroprotected against hepatitis B
Biological: Havrix — Havrix will be administered to subjects who are seronegative for anti-HAV antibodies

SUMMARY:
This study will evaluate the persistence of the immune response to HAV (Hepatitis A Virus) antigens and HBs (Hepatitis B surface) antigens in healthy adults previously vaccinated with GlaxoSmithKline (GSK) Biologicals' Twinrix Adult. The subjects will be invited for blood sampling 16, 17, 18, 19 and 20 years after vaccination to evaluate the antibody persistence. For subjects in whom low circulating antibodies are detected, the presence of immune memory against hepatitis A & B antigens will be investigated by the administration of a challenge dose of the appropriate vaccine (Havrix and/or Engerix-B) at the next planned visit.

No new subjects will be recruited during this study.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at entry into each of the long-term follow-up visits:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female who received the complete primary vaccination course in the primary study Hepatitis A and B vaccine (HAB), HAB-028 (208127/021).
* Written informed consent obtained from the subject.

All subjects must satisfy the following criteria at entry into the challenge dose phase:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female who received the complete primary vaccination course in the primary study HAB-028 (208127/021).
* Written informed consent obtained from the subject.
* Subjects who participated in the long-term follow-up (LTFU) phase of the HAB-028 (208127/021) study and for whom the antibody concentrations were below the cut-off at the last available follow-up time-point.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception for two months after the administration of the challenge dose.

Exclusion Criteria:

The following criteria should be checked before entry into each of the long-term follow-up visits. If any exclusion criterion applies, the subject must not be included in the study:

* Use of any investigational or non-registered product within 30 days prior to blood sampling.
* Administration of a hepatitis A, hepatitis B or combined hepatitis A and B vaccine outside the study procedures, since the primary study HAB-028 (208127/021).
* History of hepatitis A or hepatitis B infection since the primary study HAB-028 (208127/021).
* Administration of hepatitis A or hepatitis B immunoglobulins and/or any blood products within three months prior to blood sampling.

The following criteria should be checked before the challenge dose is administered. If any apply, the subject must not be included in the challenge dose phase:

* Use of any investigational or non-registered product within 30 days prior to study start or planned use during the study.
* Administration of a hepatitis A, hepatitis B or combined hepatitis A and B vaccine between the last LTFU visit and the challenge dose visit.
* History of hepatitis A or hepatitis B infection between the last LTFU visit and the challenge dose visit.
* History of anaphylactic reactions following the administration of vaccines.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Acute disease and/or fever at the time of enrolment.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11-06; Primary Completion 2014-07-25 (Actual); Study Completion 2014-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Agrawal A, Kolhapure S, Andani A, Ota MOC, Badur S, Karkada N, Mitra M. Long-Term Persistence of Antibody Response with Two Doses of Inactivated Hepatitis A Vaccine in Children. Infect Dis Ther. 2020 Dec;9(4):785-796. doi: 10.1007/s40121-020-00311-8. Epub 2020 Jul 24. PMID 32710245
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112267 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112267 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112267 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112267 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112267 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112267 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112267 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who entered the study at Years 16, 17, 18, 19 and 20 time points were subjects who completed the primary study and who returned for blood sampling at the considered time point. At Year 19 time point, one subject was given a challenge dose of Engerix.
Period: Year 16
Arm/Group | Twinrix Group
Started | 40
Completed | 40
Not Completed | 0
Period: Year 17
Arm/Group | Twinrix Group
Started | 32
Completed | 32
Not Completed | 0
Period: Year 18
Arm/Group | Twinrix Group
Started | 29
Completed | 29
Not Completed | 0
Period: Year 19
Arm/Group | Twinrix Group
Started | 28
Completed | 28
Not Completed | 0
Period: Year 20
Arm/Group | Twinrix Group
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Twinrix Group
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 16 Population: Number of participants at year 16 are equal to the overall number of participants analyzed, which represents the highest number of participants from year 16 to year 20.
  Years | 35.5 (2.87)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 17 Population: Number of participants analyzed represents all subjects who returned at the year 17 annual time point.
  Years
    number analyzed (Participants) | 32
    (all) | 36.3 (1.52)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 18 Population: Number of participants analyzed represents all subjects who returned at the year 18 annual time point.
  Years
    number analyzed (Participants) | 29
    (all) | 37.7 (3.25)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 19 Population: Number of participants analyzed represents all subjects who returned at the year 19 annual time point.
  Years
    number analyzed (Participants) | 28
    (all) | 38.8 (3.31)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 20 Population: Number of participants analyzed represents all subjects who returned at the year 20 annual time point.
  Years
    number analyzed (Participants) | 28
    (all) | 39.6 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 16 Population: Number of participants at year 16 are equal to the overall number of participants analyzed, which represents the highest number of participants from year 16 to year 20.
  Participants
    Female | 29
    Male | 11
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 17 Population: Number of participants analyzed represents all subjects who returned at the year 17 annual time point.
  Participants
    number analyzed (Participants) | 32
    Female | 25
    Male | 7
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 18 Population: Number of participants analyzed represents all subjects who returned at the year 18 annual time point.
  Participants
    number analyzed (Participants) | 29
    Female | 22
    Male | 7
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 19 Population: Number of participants analyzed represents all subjects who returned at the year 19 annual time point.
  Participants
    number analyzed (Participants) | 28
    Female | 21
    Male | 7
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 20 Population: Number of participants analyzed represents all subjects who returned at the year 20 annual time point.
  Participants
    number analyzed (Participants) | 28
    Female | 23
    Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seropositive for Anti-hepatitis A Virus Antibodies (Anti-HAV) and Anti-hepatitis B Surface Antigen (Anti-HBs) Antibodies and With Anti-HBs Antibody Concentrations >= 10 Milliinternational Units Per Milliliter (mIU/mL)
Description: Seropositivity for anti-HAV antibodies is defined as antibody concentrations >= 15 milliinternational units per milliliter (mIU/mL). Seropositivity for anti-HBs antibodies is defined as antibody concentrations >= 6.2 mIU/mL.
Time Frame: At Years 16, 17, 18, 19 and 20.
Population: The analysis was performed on the Long-Term (LT) According-to-Protocol (ATP) cohort for analysis of immunogenicity. They were included in the ATP analysis for the primary study, did not receive hepatitis A or B (hep A/B) vaccination that was not specified in the protocol and were not eliminated for abnormal increase of antibody concentrations.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 23
Subjects
  Anti-HAV >=15 mIU/mL [at Year 16] (N=23) | 23
  anti-HBs >= 6.2 mIU/mL [at Year 16] (N=23) | 20
  anti-HBs >= 10 mIU/mL [at Year 16] (N=23) | 20
  anti-HAV >= 15 mIU/mL [at Year 17] (N=19) | 19
  anti-HBs >= 6.2 mIU/mL [at Year 17] (N=19) | 17
  anti-HBs >= 10 mIU/mL [at Year 17] (N=19) | 17
  anti-HAV >= 15 mIU/mL [at Year 18] (N=10) | 10
  anti-HBs >= 6.2 mIU/mL [at Year 18] (N=10) | 9
  anti-HBs >= 10 mIU/mL [at Year 18] (N=10) | 9
  anti-HAV >= 15 mIU/mL [at Year 19] (N=17) | 17
  anti-HBs >= 6.2 mIU/mL [at Year 19] (N=18) | 17
  anti-HBs >= 10 mIU/mL [at Year 19] (N=18) | 17
  anti-HAV >= 15 mIU/mL [at Year 20] (N=18) | 18
  anti-HBs >= 6.2 mIU/mL [at Year 20] (N=18) | 17
  anti-HBs >= 10 mIU/mL [at Year 20] (N=18) | 17

2. Primary Outcome: Anti-HAV and Anti-HBs Geometric Mean Concentrations (GMCs)
Description: Concentrations were expressed as GMCs in mIU/mL.
Time Frame: At Years 16, 17, 18, 19 and 20.
Population: The analysis was performed on the Long-Term (LT) According-to-Protocol (ATP) cohort for analysis of immunogenicity.They were included in the ATP analysis for the primary study, did not receive hepatitis A or B vaccination that was not specified in the protocol and were not eliminated for abnormal increase of antibody concentrations.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Twinrix Group
Number analyzed (Participants) | 23
milli-international units per milliliter
  anti-HAV [at Year 16] (N=23) | 614.2 [404.1 to 933.6]
  anti-HBs [at Year 16] (N=23) | 138.7 [61.3 to 313.7]
  anti-HAV [at Year 17] (N=19) | 479.2 [298.2 to 769.9]
  anti-HBs [at Year 17] (N=19) | 165.1 [64.8 to 420.7]
  anti-HAV [at Year 18] (N=10) | 653.2 [333.2 to 1280.6]
  anti-HBs [at Year 18] (N=10) | 278.3 [70.3 to 1101.3]
  anti-HAV [at Year 19] (N=17) | 728.7 [469.6 to 1130.5]
  anti-HBs [at Year 19] (N=18) | 198.4 [80.1 to 491.3]
  anti-HAV [at Year 20] (N=18) | 511.9 [343.8 to 762.0]
  anti-HBs [at Year 20] (N=18) | 195.8 [79.9 to 480.0]

3. Secondary Outcome: Number of Subjects With Immune Response to the Challenge Vaccine Antigen
Description: None of the subjects received a challenge dose at Years 16, 17, 18 and 20 while, one subject received the challenge dose at Year 19.
Time Frame: Before, 14 days and one month after the challenge dose at Year 19.
Population: The analysis was performed on LT Total cohort that included all subjects who returned at each annual time point and who belonged to the Total Vaccinated cohort in the primary study.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
Subjects | 1

4. Secondary Outcome: Anti-hepatitis B Virus (Anti-HBs) Antibody Concentration
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) expressed as mIU/mL.
Time Frame: At Year 18, 14 days and 30 days post challenge dose (Year 19).
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
milli-international units per milliliter
  [Subject 1; at year 18] | 13.26 [NA to NA] — One subject received the challenge dose at Year 19.
  [Subject 1; 14 days post challenge dose] | 21926.00 [NA to NA] — One subject received the challenge dose at Year 19.
  [Subject 1; 30 days post challenge dose] | 12736.00 [NA to NA] — One subject received the challenge dose at Year 19.

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An unsolicited AE was defined as any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0 to 30) period after administration of the challenge dose at Year 19.
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
Subjects | 1

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 31-day (Day 0 to 30) period after administration of the challenge dose at Year 19.
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
Subjects | 0

7. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: A serious adverse event is any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, or was a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Up to Year 20.
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 40
Subjects | 0

ADVERSE EVENTS:
Time Frame: SAEs: During the 31-day (Days 0 to 30) follow-up period after the challenge dose and from the beginning of the long term follow-up to Year 20; Unsolicited symptoms: During the 31-day (Days 0 to 30) follow-up period after the challenge dose.
Description: As no challenge dose was administered during Years 16, 17, 18 and 20 time points, SAEs and other adverse events were not assessed. 1 subject received the challenge dose at Year 19 for whom the SAEs and other adverse events were assessed during the 31 day period post challenge dose. SAEs were also collected for the entire safety follow-up.
Arm/Group | Twinrix Group
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Twinrix Group (N=1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/ml). The table shows updated results following partial or complete retesting/reanalysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.